CLINICAL TRIAL: NCT02631122
Title: Ultrasound Guided Supraclavicular Brachial Plexus Block vs Retroclavicular Brachial Plexus Block: Comparison of Impact on Ipsilateral Diaphragmatic Function
Brief Title: Supraclavicular Block vs Retroclavicular Block: Incidence of Phrenic Nerve Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kamen Vlassakov, Director of Regional and Orthopedic Anesthesiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P001537
Record Dates: First submitted 2015-12-04; First posted 2015-12-16 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Phrenic Nerve Paralysis
Keywords: Retroclavicular; Supraclavicular; Diagphram; hemiparesis; nerve block; regional anesthesia; anesthesiology
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular BPNB (Active Comparator): Patients in this group will be randomized to receive an Ultrasound Guided Supraclavicular Brachial Plexus Nerve Block and outcomes will be measured over the perioperative and 1day time period.
  Interventions: Procedure: Supraclavicular vs Retroclavicular Nerve Block
- Retroclavicular BNPB (Active Comparator): Patients in this group will be randomized to receive an Ultrasound Guided Retroclavicular Brachial Plexus Nerve Block and outcomes will be measured over the perioperative and 1day time period.
  Interventions: Procedure: Supraclavicular vs Retroclavicular Nerve Block

INTERVENTIONS:
Procedure: Supraclavicular vs Retroclavicular Nerve Block — An ultrasound-guided supraclavicular or retroclavicular nerve block with 30 ml of 0.5% ropivicaine will be performed on patients scheduled for lower arm surgery; 25 ml to be delivered to the brachial plexus and 5 ml to the intercostal nerve

SUMMARY:
The aim of this study is to evaluate differences between ultrasound guided supraclavicular versus retroclavicular brachial plexus blocks: two similar brachial plexus nerve block techniques that differ in their needle trajectory and injection site.

DETAILED DESCRIPTION:
To date, there has not been a study that has compared clinically the retroclavicular brachial plexus block to the supraclavicular brachial plexus block or other brachial plexus blocks. The aim of this study is to evaluate differences between ultrasound guided supraclavicular versus retroclavicular brachial plexus blocks, with primary focus on the incidence of diminished ipsilateral hemidiaphramatic excursion (ipsilateral phrenic nerve blockade). We will also evaluate differences between the two techniques in the success of producing surgical anesthesia, procedural time to perform the block (including imaging time and needling time), block onset time, ease of quality ultrasound needle visualization, and incidence of paresthesias, vascular puncture and pneumothorax. Lastly, we will observe and compare the distribution of motor and sensory blockade of the two techniques

ELIGIBILITY:
Inclusion Criteria:

1. patients scheduled for lower arm surgery
2. patients aged 18 years or older
3. patients ASA class I-III

Exclusion Criteria:

1. Patients unable to cooperate or consent to the study
2. pre-existing neuropathy
3. significant pulmonary disease
4. contralateral phrenic nerve or diaphragmatic dysfunction
5. allergy to local anesthetics
6. infection at needle insertion site
7. history of coagulopathy
8. BMI > 40 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of IIpsilateral Diaphragmatic Paresis | 30 minutes post block, then postoperatively
  As evidence by ipsilater diagphragmatic excursion measured by Mmode ultrasound

SECONDARY OUTCOMES:
Anesthetic and analgesic efficacy | 30 minutes post block, then postoperatively
  Block success will be defined as onset of acceptable sensory and motor blockade
Procedural times (imaging time and needling time), onset time, ease of placement, and block duration | at the time of block
  Ultrasonographic block imaging times (time between ultrasound probe placement on the patient and satisfactory image of target anatomy acquisition. needling time (time between needle insertion into the skin and the end of local anesthetic injection through the block needle), onset and duration of sensory block, and proceduralist's rating of ease of block performance will be measured.
Complication rates | 1 day
  Rates of vascular puncture, pneumothorax and paresthesias will be recorded
Nerve block distribution | 30 minutes post block
  measured through sensation (cold and pin prick) over dermatomes of the brachial plexus

CONTACTS AND LOCATIONS:
Overall Officials: Kamen Vlassakov, MD, Principal Investigator — kvlassakov@partners.org
Locations (1):
- Kamen Vlassakov, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Georgiadis PL, Vlassakov KV, Patton ME, Lirk PB, Janfaza DR, Zeballos JL, Quaye AN, Patel V, Schreiber KL. Ultrasound-guided supraclavicular vs. retroclavicular block of the brachial plexus: comparison of ipsilateral diaphragmatic function: A randomised clinical trial. Eur J Anaesthesiol. 2021 Jan;38(1):64-72. doi: 10.1097/EJA.0000000000001305. PMID 32925256